CLINICAL TRIAL: NCT03958071
Title: Characteristics of IPF Patients Initiating Nintedanib, Pirfenidone or no Antifibrotic Treatment in the US
Brief Title: A Study Based on Medical Records That Looks at the Characteristics of Idiopathic Pulmonary Fibrosis Patients Grouped by the Type of Medication They Are Taking
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1199-0375
Record Dates: First submitted 2019-05-20; First posted 2019-05-21 (Actual); Results first posted 2020-12-17 (Actual); Last update posted 2021-11-15 (Actual); Status verified 2021-11

CONDITIONS: Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis | interventions — nintedanib; pirfenidone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Subjects with Idiopathic Pulmonary Fibrosis
  Interventions: Drug: Nintedanib; Drug: Pirfenidone; Other: Untreated Cohort

INTERVENTIONS:
Drug: Nintedanib — Nintedanib initiators
Drug: Pirfenidone — Pirfenidone initiators
Other: Untreated Cohort — Untreated

SUMMARY:
To understand differences in characteristics of Idiopathic Pulmonary Fibrosis (IPF) patients who are prescribed nintedanib compared to those who are prescribed pirfenidone.

ELIGIBILITY:
Inclusion Criteria:

* With ≥ 1 diagnosis for IPF (the International Classification of Diseases, Ninth Revision, Clinical Modification [ICD-9-CM] codes 516.3, 516.31, 515, or ICD-10-CM codes J84.112) in the EMR between October 1, 2013 to April 30, 2018
* With ≥ 1 prescription for nintedanib between October 1, 2014 and April 30, 2018 (the selection window)
* The date of the first prescription will be defined as the index date
* With ≥ 1 record in the EMR database during the 12 months prior to the index date (the pre-index period)
* With ≥ 1 diagnosis of IPF during the 12 months prior to the index date
* Age ≥ 40 on the index date
* IQVIA will explore also requiring ≥ 1 chest CT scan before first IPF diagnosis during the pre-index period

Exclusion Criteria:

* With ≥ 1 diagnosis of other known causes of interstitial lung disease (ILD) on the date of or after the first IPF diagnosis during the pre-index period
* Other known causes of ILD include conditions such as systemic sclerosis, rheumatoid arthritis, systemic lupus erythematosus, dermatomyositis, polymyositis, Sjögren disease, and hypersensitivity pneumonitis (ICD-9-CM codes 135, 237.7, 272.7, 277.3, 277.8, 446.21, 446.4, 495, 500-505, 506.4, 508.1, 508.8, 516.0, 516.1, 516.32-516.37, 516.2, 516.8, 516.9, 517.0, 517.2, 517.8, 518.3, 555, 710.0, 710.0-710.4, 714.0, 714.81, 720, and 759.5, or ICD-10-CM equivalent codes)
* With ≥ 1 prescription for nintedanib prior to the index date
* With ≥ 1 prescription for pirfenidone prior to or on the index date

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of the following three mutually exclusive cohorts:
  1. Nintedanib initiators, consisting of adult IPF patients who newly initiated nintedanib treatment
  2. Pirfenidone initiators, consisting of adult IPF patients who newly initiated pirfenidone treatment
  3. Untreated cohort, consisting of adult IPF patients without any prescription for antifibrotic treatment (i.e., no prescription for nintedanib nor pirfenidone)
Sampling Method: Non-Probability Sample
Enrollment: 13264 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-05-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Plymouth Meeting, Plymouth, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents, except for the following exclusions:
  1. studies in products where Boehringer Ingelheim is not the license holder;
  2. studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials;
  3. studies conducted in a single center or targeting rare diseases (because of limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datasharing

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This retrospective database study was conducted to understand differences in characteristics of Idiopathic pulmonary fibrosis (IPF) patients who were newly prescribed pirfenidone or nintedanib, and those who did not receive a prescription for an antifibrotic treatment.
Pre-assignment Details: The study includes all patients with an Idiopathic pulmonary fibrosis (IPF) diagnosis from Oct 1, 2013 to Oct 31, 2018. Data derived from IQVIA's GE Centricity EMR (Electronic medical records) data.
Groups:
- Nintedanib: Cohort of patients with an Idiopathic pulmonary fibrosis (IPF) diagnosis who were first prescribed Nintedanib from October 1, 2014 to October 31, 2018. Data derived from IQVIA's GE Centricity EMR (Electronic medical records) data. The EMR consisted of patient data from ambulatory care records in the US, representing the US population receiving healthcare in the ambulatory setting. The index date was the date of the first Nintedanib prescription.
- Pirfenidone: Cohort of patients with an Idiopathic pulmonary fibrosis (IPF) diagnosis who were first prescribed Pirfenidone from October 1, 2014 to October 31, 2018. Data derived from IQVIA's GE Centricity EMR (Electronic medical records) data. The EMR consisted of patient data from ambulatory care records in the US, representing the US population receiving healthcare in the ambulatory setting. The index date was the date of the first Pirfenidone prescription.
- Untreated: Cohort of patients with an Idiopathic pulmonary fibrosis (IPF) diagnosis who were not prescribed antifibrotic treatment (i.e., no prescription for nintedanib nor pirfenidone during the data window) from October 1, 2014 to October 31, 2018. Data derived from IQVIA's GE Centricity EMR (Electronic medical records) data. The EMR consisted of patient data from ambulatory care records in the US, representing the US population receiving healthcare in the ambulatory setting. The index date for the untreated cohort was randomly assigned to mimic the distribution of time from the earliest IPF diagnosis to index in the two treatment cohorts.
Period: Overall Study
Arm/Group | Nintedanib | Pirfenidone | Untreated
Started | 347 | 423 | 12494
Completed | 347 | 423 | 12494
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Includes all patients with an Idiopathic pulmonary fibrosis (IPF) diagnosis from Oct 1, 2013 to Oct 31, 2018. Data derived from IQVIA's GE Centricity EMR (Electronic medical records) data. The EMR consisted of patient data from ambulatory care records in the US, representing the US population receiving healthcare in the ambulatory setting.
Groups:
- Total: Total of all reporting groups
Arm/Group | Nintedanib | Pirfenidone | Untreated | Total
Number analyzed (Participants) | 347 | 423 | 12494 | 13264
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.6 (6.7) | 72.1 (6.8) | 70.9 (8.9) | 70.96 (8.79)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 234 | 281 | 6179 | 6694
  Female | 113 | 142 | 6314 | 6569
  Unknown | 0 | 0 | 1 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 305 | 370 | 10039 | 10714
  Non-white | 16 | 15 | 1093 | 1124
  Unknown | 26 | 38 | 1362 | 1426

OUTCOME MEASURES:

1. Primary Outcome: Baseline Patient Characteristics: Age
Description: IQVIA's GE Centricity Electronic medical records database was used for this study. This is an anonymized Health Insurance Portability and Accountability Act of 1996 (HIPPA) compliant database populated with patient data from ambulatory care records.
  The patient characteristic age for Idiopathic Pulmonary Fibrosis (IPF) patients at 12-month pre-treatment (baseline) was compared between each of the cohorts (nintedanib vs. pirfenidone, nintedanib vs. untreated, pirfenidone vs. untreated), differences are presented in absolute standardized differences (ASD), differences were tested using t-test for means of continuous variables, Wilcoxon signed tank test for medians of continuous variables, and Chi-square test for categorical variables.
Time Frame: Baseline characteristics were recorded 12 months pre-index event (pre-treatment).
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: years
Arm/Group | Nintedanib | Pirfenidone | Untreated
Number analyzed (Participants) | 347 | 423 | 12494
years | 71.6 (6.7) | 72.1 (6.8) | 70.9 (8.9)
Statistical Analysis 1: Comparison: Nintedanib vs Pirfenidone; Test type: Other; p = 0.2810, t-test, 2 sided; Absolute standardized differences (ASD) = -0.1027 — ASD=(X1-X2)/sqrt((s1^2+s2^2)/2). Where X denotes sample means in each cohort, and s denotes sample variances
Statistical Analysis 2: Comparison: Nintedanib vs Untreated; Test type: Other; p = 0.1421, t-test, 2 sided; Absolute standardized differences (ASD) = -0.0780 — ASD=(X1-X2)/sqrt((s1^2+s2^2)/2). Where X denotes sample means in each cohort, and s denotes sample variances
Statistical Analysis 3: Comparison: Pirfenidone vs Untreated; Test type: Other; p = 0.0048, t-test, 2 sided; Absolute standardized differences (ASD) = 0.0159 — ASD=(X1-X2)/sqrt((s1^2+s2^2)/2). Where X denotes sample means in each cohort, and s denotes sample variances

2. Secondary Outcome: Odds Ratio of Receiving Treatment (Nintedanib or Pirfenidone) vs no Treatment
Description: Odds ratio of receiving nintedanib or pirfenidone vs. no antifibrotic treatment, adjusting for patient characteristics; to identify baseline characteristics that drive initiation of a treatment while minimizing prescription bias.
  Logistic regression models were developed to assess the odds. Baseline patient characteristics that were sufficiently populated, had ASD >10% or p-value <0.05, and were agreed upon as important variables to include, were included as covariates for a full model. Linearity of age was confirmed before including it as a continuous variable in one version of the model. Backward selection was applied to develop a reduced model, only retaining covariates with p<0.1 after forcing age at index, gender, geographic region, BMI, CCI, and Chronic obstructive pulmonary disease (COPD) into the model.
  Odds presented for key patient characteristics. Odd ratio of >1 indicates increased odds of receiving treatment.
Time Frame: Baseline characteristics were recorded 12 months pre-index event (pre-treatment).
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Odds ratio
Groups:
- Overall Population: Patients with an Idiopathic pulmonary fibrosis (IPF) diagnosis who were not prescribed antifibrotic treatment, first prescribed Nintedanib or first prescribed Pirfenidone from October 1, 2014 to October 31, 2018. Data derived from IQVIA's GE Centricity EMR (Electronic medical records) data. The EMR consisted of patient data from ambulatory care records in the US, representing the US population receiving healthcare in the ambulatory setting. The index date was the date of the first Nintedanib prescription.
Arm/Group | Overall Population
Number analyzed (Participants) | 13264
Odds ratio
  Age | 1.022 [1.012 to 1.032]
  Gender | 0.490 [0.419 to 0.574]
  BMI category: Overweight | 1.359 [1.113 to 1.660]
  BMI category: Obese | 1.833 [1.483 to 2.265]
  BMI category: Very obese | 1.638 [1.281 to 2.096]
  Comorbidities: COPD | 0.581 [0.457 to 0.739]
  Comorbidities: Heart failure | 0.449 [0.299 to 0.675]
  Comorbidities: Stroke | 0.449 [0.226 to 0.889]
  Comorbidities: Hypertension | 0.663 [0.527 to 0.835]
  Comorbidities: Peripheral arterial diseases | 0.383 [0.186 to 0.787]
  Comorbidities: Severe diseases | 0.463 [0.328 to 0.653]
  Gastroesophageal reflux disease | 1.621 [1.291 to 2.036]

3. Primary Outcome: Baseline Patient Characteristics: Sex
Description: IQVIA's GE Centricity Electronic medical records database was used for this study. This is an anonymized Health Insurance Portability and Accountability Act of 1996 (HIPPA) compliant database populated with patient data from ambulatory care records.
  The patient characteristic sex for Idiopathic Pulmonary Fibrosis (IPF) patients at 12-month pre-treatment (baseline) was compared between each of the cohorts (nintedanib vs. pirfenidone, nintedanib vs. untreated, pirfenidone vs. untreated), differences are presented in absolute standardized differences (ASD), differences were tested using t-test for means of continuous variables, Wilcoxon signed tank test for medians of continuous variables, and Chi-square test for categorical variables.
Time Frame: Baseline characteristics were recorded 12 months pre-index event (pre-treatment).
Population: Includes all patients with an Idiopathic pulmonary fibrosis (IPF) diagnosis from Oct 1, 2013 to Oct 31, 2018. Data derived from IQVIA's GE Centricity EMR (Electronic medical records) data. The EMR consisted of patient data from ambulatory care records in the US, representing the US population receiving healthcare in the ambulatory setting. One patient from the untreated cohort was missing gender information and is not shown in the table
Measure: Count of Participants; unit: Participants
Arm/Group | Nintedanib | Pirfenidone | Untreated
Number analyzed (Participants) | 347 | 423 | 12493
Participants
  Male | 234 | 281 | 6179
  Female | 113 | 142 | 6314
Statistical Analysis 1: Comparison: Nintedanib vs Pirfenidone; Test type: Other; p = 0.7681, Chi-squared; Absolute standardized differences (ASD) = 0.0214 — ASD=(p1-p2)/(sqrt(p1^(1-p1)+p2(1-p2))/2). Where p denotes proportion of a binary variable in each cohort
Statistical Analysis 2: Comparison: Nintedanib vs Untreated; Test type: Other; p < .0001, Chi-squared; Absolute standardized differences (ASD) = 0.3710 — ASD=(p1-p2)/(sqrt(p1^(1-p1)+p2(1-p2))/2). Where p denotes proportion of a binary variable in each cohort
Statistical Analysis 3: Comparison: Pirfenidone vs Untreated; Test type: Other; p < .0001, Chi-squared; Absolute standardized differences (ASD) = 0.3490 — ASD=(p1-p2)/(sqrt(p1^(1-p1)+p2(1-p2))/2). Where p denotes proportion of a binary variable in each cohort

4. Primary Outcome: Baseline Patient Characteristics: BMI
Description: The patient characteristic Body mass index (BMI) for Idiopathic Pulmonary Fibrosis (IPF) patients at 12-month pre-treatment (baseline) was compared between each of the cohorts (nintedanib vs. pirfenidone, nintedanib vs. untreated, pirfenidone vs. untreated), differences are presented in absolute standardized differences (ASD), differences were tested using t-test for means of continuous variables, Wilcoxon signed tank test for medians of continuous variables, and Chi-square test for categorical variables.
Time Frame: Baseline characteristics were recorded 12 months pre-index event (pre-treatment).
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: kilogram/height in meters squared(kg/m²)
Arm/Group | Nintedanib | Pirfenidone | Untreated
Number analyzed (Participants) | 347 | 423 | 12494
kilogram/height in meters squared(kg/m²) | 29.5 (6.4) | 30.1 (5.8) | 28.6 (6.5)
Statistical Analysis 1: Comparison: Nintedanib vs Pirfenidone; Test type: Other; p = 0.1659, t-test, 2 sided; Absolute standardized differences (ASD) = -0.1257 — ASD=(X1-X2)/sqrt((s1^2+s2^2)/2). Where X denotes sample means in each cohort, and s denotes sample variances
Statistical Analysis 2: Comparison: Nintedanib vs Untreated; Test type: Other; p = 0.0112, t-test, 2 sided; Absolute standardized differences (ASD) = 0.1566 — ASD=(X1-X2)/sqrt((s1^2+s2^2)/2). Where X denotes sample means in each cohort, and s denotes sample variances
Statistical Analysis 3: Comparison: Pirfenidone vs Untreated; Test type: Other; p < .0001, t-test, 2 sided; Absolute standardized differences (ASD) = 0.3019 — ASD=(X1-X2)/sqrt((s1^2+s2^2)/2). Where X denotes sample means in each cohort, and s denotes sample variances

5. Primary Outcome: Baseline Patient Characteristics: Charlson Comorbidity Index (CCI)
Description: IQVIA's GE Centricity Electronic medical records database was used for this study. This is an anonymized HIPPA compliant database populated with patient data from ambulatory care records. Charlson Comorbidity Index (CCI) for Idiopathic Pulmonary Fibrosis (IPF) patients at 12-month pre-treatment (baseline) was compared between each of the cohorts.
  The Charlson Comorbidity Index is a method of categorizing comorbidities of patients based on the International Classification of Diseases (ICD) diagnosis. Each comorbidity category has an associated weight (from 1 to 6), based on the adjusted risk of mortality or resource use, and the sum of all the weights results in a single comorbidity score for a patient. A score of zero indicates that no comorbidities were found. The higher the score, the more likely the predicted outcome will result in mortality or higher resource use. Up to 12 comorbidities with various weightings can result in a maximum score of 24. The minimum score is zero.
Time Frame: Baseline characteristics were recorded 12 months pre-index event (pre-treatment).
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Nintedanib | Pirfenidone | Untreated
Number analyzed (Participants) | 347 | 423 | 12494
Score on a scale | 0.71 (1.0) | 0.79 (1.1) | 1.09 (1.4)
Statistical Analysis 1: Comparison: Nintedanib vs Pirfenidone; Test type: Other; p = 0.3260, t-test, 2 sided; Absolute standardized differences (ASD) = -0.0209 — ASD=(X1-X2)/sqrt((s1^2+s2^2)/2). Where X denotes sample means in each cohort, and s denotes sample variances
Statistical Analysis 2: Comparison: Nintedanib vs Untreated; Test type: Other; p < .0001, t-test, 2 sided; Absolute standardized differences (ASD) = -0.2694 — ASD=(X1-X2)/sqrt((s1^2+s2^2)/2). Where X denotes sample means in each cohort, and s denotes sample variances
Statistical Analysis 3: Comparison: Pirfenidone vs Untreated; Test type: Other; p < .0001, t-test, 2 sided; Absolute standardized differences (ASD) = -0.2352 — ASD=(X1-X2)/sqrt((s1^2+s2^2)/2). Where X denotes sample means in each cohort, and s denotes sample variances

6. Primary Outcome: Baseline Patient Characteristics: Number of Participants Using Inhaled Corticosteroids at Baseline
Description: IQVIA's GE Centricity Electronic medical records database was used for this study. This is an anonymized Health Insurance Portability and Accountability Act of 1996 (HIPPA) compliant database populated with patient data from ambulatory care records.
  Treatment with inhaled corticosteroids for Idiopathic Pulmonary Fibrosis (IPF) patients at 12-month pre-treatment (baseline) was compared between each of the cohorts (nintedanib vs. pirfenidone, nintedanib vs. untreated, pirfenidone vs. untreated), differences are presented in absolute standardized differences (ASD), differences were tested using t-test for means of continuous variables, Wilcoxon signed tank test for medians of continuous variables, and Chi-square test for categorical variables.
Time Frame: Baseline characteristics were recorded 12 months pre-index event (pre-treatment).
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Nintedanib | Pirfenidone | Untreated
Number analyzed (Participants) | 347 | 423 | 12494
Participants | 125 | 134 | 3311
Statistical Analysis 1: Comparison: Nintedanib vs Pirfenidone; Test type: Other; p = 0.2042, Chi-squared; Absolute standardized differences (ASD) = 0.09 — ASD=(p1-p2)/(sqrt(p1^(1-p1)+p2(1-p2))/2). Where p denotes proportion of a binary variable in each cohort
Statistical Analysis 2: Comparison: Nintedanib vs Untreated; Test type: Other; p < .0001, Chi-squared; Absolute standardized differences (ASD) = 0.21 — ASD=(p1-p2)/(sqrt(p1^(1-p1)+p2(1-p2))/2). Where p denotes proportion of a binary variable in each cohort
Statistical Analysis 3: Comparison: Pirfenidone vs Untreated; Test type: Other; p = 0.02, Chi-squared; Absolute standardized differences (ASD) = 0.11 — ASD=(p1-p2)/(sqrt(p1^(1-p1)+p2(1-p2))/2). Where p denotes proportion of a binary variable in each cohort

7. Primary Outcome: Baseline Patient Characteristics: Number of Participants Using Proton Pump Inhibitors at Baseline
Description: IQVIA's GE Centricity Electronic medical records database was used for this study. This is an anonymized Health Insurance Portability and Accountability Act of 1996 (HIPPA) compliant database populated with patient data from ambulatory care records.
  Treatment with Proton pump inhibitors for Idiopathic Pulmonary Fibrosis (IPF) patients at 12-month pre-treatment (baseline) was compared between each of the cohorts (nintedanib vs. pirfenidone, nintedanib vs. untreated, pirfenidone vs. untreated), differences are presented in absolute standardized differences (ASD), differences were tested using t-test for means of continuous variables, Wilcoxon signed tank test for medians of continuous variables, and Chi-square test for categorical variables.
Time Frame: Baseline characteristics were recorded 12 months pre-index event (pre-treatment).
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Nintedanib | Pirfenidone | Untreated
Number analyzed (Participants) | 347 | 423 | 12494
Participants | 113 | 133 | 3141
Statistical Analysis 1: Comparison: Nintedanib vs Pirfenidone; Test type: Other; p = 0.7395, Chi-squared; Absolute standardized differences (ASD) = 0.0241 — ASD=(p1-p2)/(sqrt(p1^(1-p1)+p2(1-p2))/2). Where p denotes proportion of a binary variable in each cohort
Statistical Analysis 2: Comparison: Nintedanib vs Untreated; Test type: Other; p = 0.0017, Chi-squared; Absolute standardized differences (ASD) = 0.1644 — ASD=(p1-p2)/(sqrt(p1^(1-p1)+p2(1-p2))/2). Where p denotes proportion of a binary variable in each cohort
Statistical Analysis 3: Comparison: Pirfenidone vs Untreated; Test type: Other; p = 0.0034, Chi-squared; Absolute standardized differences (ASD) = 0.1403 — ASD=(p1-p2)/(sqrt(p1^(1-p1)+p2(1-p2))/2). Where p denotes proportion of a binary variable in each cohort

ADVERSE EVENTS:
Description: Not applicable; the IQVIA GE Centricity EMR database is a secondary database which consists of fully de-identified data. Therefore, it is not possible to identify/report individual case safety reports. All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed.
Arm/Group | Nintedanib | Pirfenidone | Untreated
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Limitations common to retrospective database studies: high proportion of missing data and it is possible that patients who received out-of-system care and treatments were not fully captured in the data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-18): https://cdn.clinicaltrials.gov/large-docs/71/NCT03958071/Prot_SAP_000.pdf